CLINICAL TRIAL: NCT01302301
Title: Endoscopic Submucosal Tunnel Dissection for Endolumenal Partial Myotomy of the Lower Esophageal Sphincter for Atypical Primary Motility Disorders Such as Achalasia and Esophageal Spasm
Brief Title: Endolumenal Partial Myotomy for Esophageal Motility Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Oregon Clinic (Other)
Responsible Party: Lee L. Swanstrom, MD, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROV10-117A
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2010-11

CONDITIONS: Esophageal Motility Disorders
Keywords: endolumenal myotomy, per oral endoscopic myotomy
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Per oral endolumenal myotomy — flexible endoscopic submucosal esophageal partial myotomy

SUMMARY:
Achalasia and esophageal spasm are primary esophageal motility disorders where the lower esophageal sphincter fails to relax in response to swallowing with no well understood underlying cause. Surgical myotomy represents an appropriate therapeutic option. The purpose of this study is to evaluate flexible endoscopic myotomy a novel therapeutic approach to overcome the need for invasive surgery.

DETAILED DESCRIPTION:
In this study, the investigators propose the use of a recent endolumenal technique for partial myotomy in patients suffering from primary esophageal motility disorders.

Under general anesthesia patients will have upper endoscopy. Submucosal injection and mucosal incision is created for entry into the submucosal space. A submucosal tunnel is then created using a needle knife or blunt dissection as appropriate. Dissection will continue distally beyond the lower esophageal sphincter. The inner circular muscle fibers will then be divided to achieve an adequate myotomy length. The mucosal entry is then closed appropriately.

Results will be compared to historical data of conventional Heller myotomies.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for elective Heller myotomy
* Ability to undergo general anesthesia
* Ability to give informed consent

Exclusion Criteria:

* Previous mediastinal or esophageal surgery
* Contraindications for EGD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Esophageal Function Tests | 6 month
  upper endoscopy, barium swallow, esophageal manometry,ph Test

SECONDARY OUTCOMES:
Quality of life score | 6 months
  quality of life questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

REFERENCES:
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937